CLINICAL TRIAL: NCT04089553
Title: An Open-label, Multi-drug, Multi-center Phase II Combination Study of AZD4635 in Patients With Prostate Cancer
Brief Title: An Open-label, Phase II Study of AZD4635 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8731C00001; GU 156 (Other: Sarah Cannon Development Innovations, LLC); 264471 (Other: Parexel International (IRL) Limited)
Record Dates: First submitted 2019-08-29; First posted 2019-09-13 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Prostate cancer; AZD4635; oleclumab; durvalumab; MEDI9447; Adenosine 2A Receptor Antagonist; A2AR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) (Experimental): Participants will receive monotherapy of AZD4635 75 mg orally once daily (QD) for first 14 days and thereafter will continue to receive 75 mg orally QD in combination with durvalumab 1500 mg intravenously (IV) every 4 weeks (Q4W) until will derive clinical benefit as judged by the investigator, confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurs first.
  Interventions: Drug: AZD4635; Drug: Durvalumab
- Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg) (Experimental): Participants will receive combination therapy of AZD4635 (50 mg / 75 mg orally QD) and oleclumab 1500 mg IV (every 2 weeks of 28-day cycle for the first 4 doses and Q4W thereafter) until will derive clinical benefit as judged by the investigator or until confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurs first.
  Interventions: Drug: AZD4635; Drug: Oleclumab

INTERVENTIONS:
Drug: AZD4635 — In Module 1, participants will receive AZD4635 75 mg capsule orally QD for first 14 days and thereafter will continue to receive 75 mg orally QD Q4W.
  In Module 2, participants will receive AZD4635 50 mg / 75 mg capsule orally QD Q2W of 28-day cycle for the first 4 doses and Q4W thereafter.
  In both modules, participants will receive treatment until will derive clinical benefit as judged by the investigator or until confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurs first.
Drug: Oleclumab — In Module 2, participants will receive oleclumab 1500 mg IV (solution for infusion after dilution, 50 mg/mL) Q2W of 28-day cycle for the first 4 doses and Q4W thereafter until will derive clinical benefit as judged by the investigator or until confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurs first.
  Other Names: MEDI9447
  Arms: Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Drug: Durvalumab — In Module 1 after monotherapy of AZD4635, participants will receive durvalumab 1500 mg IV (solution for infusion after dilution, 50 mg/mL) Q4W until will derive clinical benefit as judged by the investigator or until confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurs first.
  Other Names: Imfinzi, MEDI4736
  Arms: Module 1 (AZD4635 75 mg + Durvalumab 1500 mg)

SUMMARY:
This is an open-label Phase II modular study in participants with prostate cancer which will assess safety, efficacy, and tolerability of AZD4635 in combination with other therapeutic agents in different treatment arms (referred to as modules).

Combinations to be studied include: 1) Module 1: AZD4635 plus durvalumab; 2) Module 2: AZD4635 plus oleclumab.

DETAILED DESCRIPTION:
This is an open-label Phase II modular study in participants with prostate cancer which will assess safety, efficacy, and tolerability of AZD4635 in combination with other therapeutic agents in different treatment arm (referred to as modules).

Combinations to be studied include: 1) Module 1: AZD4635 plus durvalumab; 2) Module 2: AZD4635 plus oleclumab.

All participants will be allocated into a module using an Interactive Web Response System (IWRS). Randomization will occur when patients meet eligibility criteria for two or more modules that are currently recruiting. If participants only meet the criteria for one currently recruiting module, they will be allocated to that module without randomization taking place.

The primary objective of the clinical study is to evaluate the efficacy of each combination therapy by: 1) assessing the objective response rate (ORR) of participants with measurable disease (response will be determined by Response Evaluation Criteria in Solid Tumours [RECIST 1.1]); 2) assessing the prostate-specific antiget (PSA) confirmed response rate of each combination therapy (PSA confirmed response rate is defined as the proportion of participants with a reduction in the PSA level of ≥50% measured from baseline to the lowest post-baseline PSA result measured twice, at least 3 weeks apart by the Prostate Cancer Working Group 3 criteria [PCWG3]).

The safety endpoints include assessment of adverse events and serious adverse events, physical examinations, vital signs, and collection of clinical chemistry/hematology parameters

There will be approximately 30 PSA evaluable participants in each module, and approximately 20 participants will have RECIST measurable disease at baseline in each module. If any of the required participants for PSA and/or ORR are not evaluable for PSA response or tumor response, respectively, they may be replaced at the sponsor's discretion.

ELIGIBILITY:
Inclusion Criteria for all Patients in all Modules:

1. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses
2. Participant must be ≥18 years of age at the time of signing the inform consent form (ICF)
3. Participants must have prostate cancer with histological or cytological confirmation
4. Participants must have previously received and progressed on standard-of-care therapy(ies)
5. Participants must be able to provide an archival tumor tissue sample. If archival tumor tissue is not available, then tissue from a fresh tumor biopsy is required.
6. All participants will be required to have a site of disease that is safely accessible for biopsy (paired) upon enrollment unless there are sufficient paired samples for the analysis. Accessible lesions are defined as those which are biopsiable (at screening) and amenable to repeat biopsy (after 2 weeks of AZD4635 therapy), unless clinically contraindicated. The provision of paired biopsies will be closely monitored to ensure the desired number of biopsiable participants are enrolled and investigators are aware of this requirement at all times.
7. Participants with measurable disease must have at least 1 documented lesion on either a bone scan or a computed tomography (CT)/ magnetic resonance imaging (MRI) scan that can be followed for response and is suitable for repeated measurement, or participants with non-measurable disease must have measurable PSA ≥1.0 ng/mL if the confirmed rise is the only indication of progression (excluding small cell carcinoma) 8 Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no clinical deterioration over the previous 2 weeks prior to the 28-day screening period and likely able to complete at least 12 weeks of treatment.

9. Ability to swallow and retain oral medication. 10. Must have life expectancy of at least 12 weeks 11. Body weight ≥ 35 kg at screening 12. Willingness to adhere to the study treatment-specific contraception requirements: Participants must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign ICF) and for 3 months after the last dose of AZD4635 to prevent pregnancy in a female partner. Male participants must not donate or bank sperm for 24 weeks after treatment.

Inclusion Criteria for Modules 1 and 2:

1. Participants must have metastatic castrate resistant prostate cancer with histological or cytological confirmation. Participant may have bone-only metastatic disease.
2. Participants must have had either orchiectomy or be on luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy with testosterone <50 ng/dL and agree to stay on LHRH agonist or antagonist therapy during the study
3. Participants must have previously received and progressed on ≥2 lines of approved systemic therapy for metastatic castration-resistant prostate cancer (mCRPC), including a second generation hormonal agent (e.g, abiraterone, enzalutamide, or apalutamide)
4. Participants must have evidence of mCRPC that progressed within 6 months prior to screening according to one of the following:

   1. PSA progression as defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each assessment, where the PSA value at screening should be ≥ 1.0 ng/mL.
   2. Radiographic disease progression in soft tissue based on RECIST Version 1.1 criteria with or without PSA progression.
   3. Radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on bone scan with or without PSA progression.

Exclusion Criteria for all Participants in all Modules:

1. History or presence of another primary invasive malignancy except for: malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of study drug and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease; localized non-invasive primary carcinoma under surveillance
2. Refractory nausea and vomiting, chronic gastrointestinal diseases, or previous significant small bowel resection that would preclude adequate absorption of AZD4635.
3. Previously untreated brain metastases. Participants who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 21 days previously and there is no evidence of central nervous system (CNS) disease progression or mild neurologic symptoms.
4. With the exception of alopecia, lymphopenia, and hypothyroidism, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) Grade 1 at the time of starting study treatment
5. Participants with prior ≥ Grade 3, serious, or life threatening immune-mediated reactions following prior anti-PD-1, anti-PD-L1, or other immuno-oncology therapies.
6. Prior history of myocardial infarction, transient ischemic attack, or stroke in the last 3 months
7. Participants must have normotensive or well controlled blood pressure (<150/90), with or without current antihypertensive treatment. If there is a diagnosis or history of hypertension, participant must have adequately controlled blood pressure on antihypertensive medications, as demonstrated by 2 blood pressure measurements taken in the clinical setting by a medical professional within 1 week prior to enrollment. Patients on a hypertensive medication must be willing and able to measure and record blood pressure readings twice-daily for a minimum of 3 weeks.
8. As judged by the Investigator or Medical Monitor, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B virus [known positive HBV surface antigen (HBsAg) result], hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies), or active hepatitis A. Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Screening for chronic conditions is not required.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis, Crohn's disease], diverticulitis, celiac disease, systemic lupus erythematous, Wegener's syndrome, myasthenia gravis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune pneumonitis, autoimmune nephritis or nephropathy, etc.) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion: a) vitiligo or alopecia, b) hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement, c) psoriasis or eczema not requiring systemic therapy for disease control, d) celiac disease controlled by diet alone.
10. Prior/concomitant therapy with AZD4635 or any other A2AR antagonist.
11. Ongoing corticosteroid use, at doses above physiologic replacement therapy. The following are exceptions to this criterion: a) use of intranasal, inhaled, topical orticosteroids, local steroid injections (e.g. intra-articular injections), b) steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication) are permitted, c) systemic corticosteroids at physiologic doses below 10 mg/day of prednisone or equivalent.
12. The following intervals between the end of the prior treatment and first dose of study drug must be observed: a) anticancer therapy: ≥21 days or 5 half-lives (whichever is shorter) of the first dose of study drug. At least 7 days must have elapsed between the last dose of such agent and the first dose of study drug. (Exception: androgen-deprivation therapy is required to maintain castrate levels of testosterone (˂50 ng/dL), b) concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
13. Major surgery (as defined by the Medical Monitor, excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
14. Minor surgical procedures (as defined by the Medical Monitor) within 7 days of the first dose of study treatment.
15. Participant is receiving medications or other products known to be sensitive breast cancer resistance protein (BCRP) or organic anion transporter polypeptide 1 (OATP1B1), OATP1B3, organic anionic transporter 1 (OAT1), organic cation transporter 1 (OCT1), OCT2, multidrug and toxin extrusion protein 1 (MATE1) and P glycoprotein (P-gp) substrates or potent or moderate inhibitors/inducers of CYP1A2, which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of AZD4635.
16. Concomitant medications with another A1R antagonist that would increase risk of seizure (e.g., theophylline, aminophylline).
17. Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
18. Ongoing treatment with Coumadin
19. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug
20. Herbal preparations/medications are not allowed throughout the study, including but not limited to: St. John's wort, kava, ephedra (ma huang), ginkgo biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Participants should stop using these herbal medications 7 days prior to the first dose of AZD4635. Exceptions may be agreed upon, but the circumstances must be reviewed by the Medical Monitor in advance.
21. Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks, of the first dose of study treatment.
22. Enrollment into another therapeutic clinical trial. (Exception: Participants are allowed to participate in investigational imaging or non-interventional studies.)
23. History of hypersensitivity to AZD4635 or drugs with a similar chemical structure or class to AZD4635.
24. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTcF) >470 msec obtained from 3 ECGs
    * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
    * Any concomitant medication with known QT interval prolongation. Participants receiving a medication(s) known to prolong the QT interval may be discussed with the Medical Monitor or Sponsor for study approval.
    * Ejection fraction <55% or the lower limit of normal of the institutional standard
25. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 x 10⁹/L
    * Platelet count <100 x 10⁹/L
    * Hemoglobin <9.0 g/dL
    * Alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Total bilirubin (TBL) >1.5 times ULN
    * Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
26. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and its representatives and/or staff at the study site).
27. Judgment by the Investigator or Medical Monitor that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
28. Participation in another clinical interventional study or if participant has already received at least one dose of study drug in the present study

Exclusion Criteria for Module 1:

1. Prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines.
2. History of active primary immunodeficiency.
3. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice)

Exclusion Criteria for Module 2:

1. Prior receipt of any immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, and anti-PD-L1 antibodies and agents targeting CD73, CD39, or adenosine receptors, excluding therapeutic anticancer vaccines.
2. Known history of allergy or reaction to any component of oleclumab formulation or history of anaphylaxis to any human gammaglobulin therapy.
3. History of venous thrombosis within the past 3 months.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will enroll only male participants because the condition being studied is metastatic castration-resistant prostate cancer.
Enrollment: 59 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2023-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Denver, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Decatur, Illinois
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Falchook GS, Reeves J, Gandhi S, Spigel DR, Arrowsmith E, George DJ, Karlix J, Pouliot G, Hattersley MM, Gangl ET, James GD, Thompson J, Russell DL, Patel B, Kumar R, Lim E. A phase 2 study of AZD4635 in combination with durvalumab or oleclumab in patients with metastatic castration-resistant prostate cancer. Cancer Immunol Immunother. 2024 Mar 2;73(4):72. doi: 10.1007/s00262-024-03640-6. PMID 38430405
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00001&attachmentIdentifier=2f03c1ac-221c-46ac-a061-a5a325386c25&fileName=D8731C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00001&attachmentIdentifier=0c352242-2780-4f98-ab98-094a9e2ea969&fileName=D8731C00001_SAP_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8731C00001&attachmentIdentifier=ed1b4676-5840-457d-a28e-bed9b1685bd8&fileName=D8731C00001_CSP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Module 1 (AZD4635 75 mg + Durvalumab 1500 mg): Participants received monotherapy of AZD4635 75 mg orally once daily (QD) for first 14 days and thereafter continued to receive 75 mg orally QD in combination with durvalumab 1500 mg intravenously (IV) every 4 weeks (Q4W) until derived clinical benefit as judged by the investigator, confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurred first.
- Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg): Participants received combination therapy of AZD4635 (50 mg / 75 mg orally QD) and oleclumab 1500 mg IV (every 2 weeks of 28-day cycle for the first 4 doses and Q4W thereafter) until derived clinical benefit as judged by the investigator or until confirmed disease progression, unacceptable toxicity, started alternative anticancer therapy, withdrawal of consent, or lost to-follow-up, whichever occurred first.
Period: Overall Study
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Started | 29 | 30
Completed (Patients ongoing study treatment at data cut-off date) | 3 | 2
Not Completed | 26 | 28
Not completed — Death | 1 | 1
Not completed — Progressive disease - objective (AZD4635) | 13 | 20
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease - subjective (AZD4635) | 6 | 3
Not completed — Other | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg) | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (7.10) | 72.7 (7.33) | 72.5 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: The confirmed objective response is defined as confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 guidelines, assessed by computed tomography (CT) scan/ magnetic resonance imaging (MRI) scan/ positron emission tomography (PET) scan and bone scan. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: Baseline (Day -28) through end of study (last participant last visit) (approximately 22 months)
Population: Tumor response analysis set included all participants who received at least one dose of study drug and had a baseline tumor assessment and measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 20 | 21
Percentage of participants | 5 [0.1 to 24.9] | 0 [NA to 16.1] — Lower limit of 95% CI was not reached because an insufficient number of participants had objective response.

2. Primary Outcome: Percentage of Participants With Confirmed Prostate-specific Antigen (PSA) Response Per Prostate Cancer Working Group 3 (PCWG3) Criteria
Description: A confirmed PSA response is defined as reduction in the PSA level of >= 50% from baseline to the lowest post-baseline PSA results, measured twice, at least 3 weeks apart by the PCWG3 criteria.
Time Frame: Baseline (Day -28) through end of study (last participant last visit) (approximately 22 months)
Population: The PSA response analysis set included all participants who received at least one dose of study drug and had an abnormal baseline PSA data (>= 1 ng/mL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 28 | 30
Percentage of participants | 3.6 [0.1 to 18.3] | 3.3 [0.1 to 17.2]

3. Secondary Outcome: Percentage of Participants With Radiological Progression Free Survival (rPFS) at 6 Months
Description: The rPFS is defined as the time interval from the first dose of AZD4635 until the date of radiological disease progression (RECIST 1.1 for soft tissue lesions and PCWG3 criteria for bone lesions) or death (by any cause in the absence of progression) regardless of whether the participant withdrew from study therapy or received another anti-cancer therapy prior to progression. The progressive disease for soft lesions per RECIST 1.1 (assessed by CT/MRI/PET scan) is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum in the study, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The progressive disease for bone lesions per PCWG3 is defined as at least 2 or more new metastatic bone lesions observed compared to baseline assessment (Day -28), with confirmation scan performed at least 6-week later.
Time Frame: Baseline (Day -28) through end of study (last participant last visit) (approximately 22 months)
Population: Efficacy analysis set included all participants who received at least one dose of study drug and had a baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 29 | 30
Percentage of participants | 8.8 [0.71 to 30.28] | 11.1 [2.83 to 25.75]

4. Secondary Outcome: Duration of Response (DoR)
Description: The DoR is defined as the time from the date of first documented response (confirmed CR/PR) until date of documented progression or death in the absence of disease progression. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression or not evaluable response in-between. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The DoR was estimated using Kaplan-Meier method.
Time Frame: Baseline (Day -28) through end of study (last participant last visit) (approximately 22 months)
Population: Tumor response analysis set included all participants who received at least one dose of study drug and had a baseline tumor assessment (Day -28) and measurable disease at baseline. Participants who had confirmed CR/PR were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 1 | 0
Months | NA [NA to NA] — Median and inter-quartile range could not be determined because insufficient number of participants were evaluated for the specified arm. |

5. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from date of first study dose until the date of death due to any cause. The median of OS was estimated using Kaplan-Meier method and CI was derived based on Brookmeyer-Crowley method.
Time Frame: Baseline (Day -28) through end of study (last participant last visit) (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 29 | 30
Months | 10.72 [7.20 to NA] — Upper limit of 95% CI was not determined because an insufficient number of participants had events. | NA [10.65 to NA] — Median and upper limit of 95% CI were not determined because an insufficient number of participants had events.

6. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to Durvalumab
Description: The detection of the immunogenicity of monoclonal antibody to durvalumab was performed using a validated immunoassay method. Participants with positive ADA to durvalumab are reported.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 4, and 7 and 90 days following the last dose of durvalumab (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of durvalumab and had at least one post dose ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg)
Number analyzed (Participants) | 26
Participants | 4

7. Secondary Outcome: Number of Participants With Positive ADA to Oleclumab
Description: The detection of the immunogenicity of monoclonal antibody to oleclumab was performed using a validated immunoassay method. Participants with positive ADA to oleclumab are reported.
Time Frame: Pre-dose on Day 1 of Cycles 1, 3, 5, and every 12 weeks thereafter, and 90 days following the last dose of oleclumab (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of oleclumab and had at least one post dose ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 24
Participants | 1

8. Secondary Outcome: Plasma Concentrations of AZD4635 and Its Metabolites (SSP-005173 and SSP-005174)
Description: Plasma concentrations of AZD4635 and its metabolites (SSP-005173 and SSP-005174) are reported.
Time Frame: Predose on Day 1 of Cycle 7
Population: Pharmacokinetics (PK) analysis set included all participants who received at least one dose of AZD4635 and had at least 1 reportable PK concentration at Cycle 7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 3 | 3
ng/mL
  AZD4635 concentration | 97.64 (21.67) | 75.47 (83.37)
  SSP-005173 concentration | 5.386 (95.48) | 6.905 (160.2)
  SSP-005174 concentration | 13.24 (69.59) | 11.79 (75.23)

9. Secondary Outcome: Plasma Concentration of Durvalumab
Description: Plasma concentration of durvalumab is reported.
Time Frame: Predose and end of infusion on Day 1 of Cycle 7
Population: The PK analysis set included all participants who received at least one dose of durvalumab and had at least 1 reportable PK concentration at Cycle 7. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg)
Number analyzed (Participants) | 2
ng/mL
  Pre-dose | NA (NA) — Geometric mean and geometric coefficient of variation were not reported as an insufficient participants were evaluated for the specified time point.
  End of infusion: number analyzed (Participants) | 1
  End of infusion | NA (NA) — Geometric mean and geometric coefficient of variation were not reported as only one participant was evaluated for the specified time point.

10. Secondary Outcome: Plasma Concentration of Oleclumab
Description: Plasma concentration of oleclumab is reported.
Time Frame: Predose and 10 minutes end of infusion on Day 1 of Cycle 14
Population: The PK analysis set included all participants who received at least one dose of oleclumab and had at least 1 reportable PK concentration at Cycle 7. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 1
mcg/mL
  Pre-dose | NA (NA) — Geometric mean and geometric coefficient of variation were not reported as only one participant was evaluated for the specified time point.
  10 minutes end of infusion | NA (NA) — Geometric mean and geometric coefficient of variation were not reported as only one participant was evaluated for the specified time point.

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 29 | 30
Participants
  Any TEAEs | 27 | 29
  Any TESAEs | 6 | 8

12. Secondary Outcome: Number of Participants With Common Terminology Criteria for Adverse Events (CTCAE) Grade Change in Laboratory Parameters From Baseline to Grade 3 or More
Description: Laboratory parameters included hematology, coagulation, clinical chemistry, and urinalysis. The CTCAE is a descriptive terminology is used for AE reporting. The CTCAE v5.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 as mild AE, Grade 2 as moderate AE, Grade 3 as severe AE, Grade 4 as life-threatening or disabling AE, and Grade 5 as death related to AE. Participants with CTCAE v5.0 grade change in laboratory parameters from baseline (Day 1 before the start of study treatment) to Grade 3 or more are reported.
Time Frame: Baseline (Day 1) through 90 days after the last dose of study drug (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 29 | 30
Participants
  Hemoglobin (low) | 2 | 2
  Leukocytes (low) | 0 | 1
  Lymphocytes (low) | 4 | 6
  Albumin | 1 | 0
  Alkaline Phosphatase | 1 | 0
  Gamma Glutamyl Transferase | 1 | 0
  Lipase | 3 | 1
  Sodium (low) | 1 | 1

13. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examination Reported as TEAEs
Description: Vital signs assessment included body temperature, respiration rate, pulse rate, blood pressure, and weight. Participants with abnormal vital signs and/or abnormal physical examination reported as TEAEs are reported.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 22 months)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
Number analyzed (Participants) | 29 | 30
Participants
  Cachexia | 1 | 1
  Hypertension | 1 | 2
  Hypotension | 0 | 1
  Gait disturbance | 0 | 1
  Pyrexia | 0 | 2

ADVERSE EVENTS:
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 22 months)
Arm/Group | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg)
All-Cause Mortality (participants affected / at risk) | 12/29 | 11/30
Serious Adverse Events (participants affected / at risk) | 6/29 | 8/30
Other Adverse Events (participants affected / at risk) | 27/29 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) (N=29) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg) (N=30)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Module 1 (AZD4635 75 mg + Durvalumab 1500 mg) (N=29) | Module 2 (AZD4635 50 / 75 mg + Oleclumab 1500 mg) (N=30)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (4)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (14) | 16 (19)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (9) | 7 (8)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 7 (7) | 13 (13)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (6)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 5 (5) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT04089553/Prot_005.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04089553/SAP_006.pdf